CLINICAL TRIAL: NCT00276822
Title: Facilitating Caring Communication for People With Cancer: The Case of Breast Cancer
Brief Title: Improving Communication With Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary findings did not support purpose.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NU 05B4; P30CA060553 (NIH); NU-05B4; NU-IRB-0608-011; STU00018976 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Other: communication intervention — Patient Education Programs to include surveys, questionnaires, interviews, and videos.

SUMMARY:
RATIONALE: An education program based on patients' health communication needs may improve patients' overall healthcare experience and sense of control.

PURPOSE: This clinical trial is studying the health communication needs of patients with breast cancer to develop patient education programs.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine patients' health communication needs during the first 6 months of care by interviewing patients with breast cancer (as well as their families, caregivers, and healthcare teams) and observing interactions between patients and oncologists throughout the trajectory of care from initial diagnosis through the initial treatment course.
* Determine patients' health communication needs at the point of bone metastases by interviewing patients with breast cancer (as well as their families, caregivers, and healthcare teams) and observing interactions between patients and oncologists in the Hematology-Oncology Clinic.
* Develop Patient Education Programs to help meet patients' health communication needs by conveying information about essential elements of cancer care in a clear and consistent manner, thus allowing clinicians to focus more attention on answering questions, engaging in counseling, and responding to emotional issues.
* Create a Patient Education Program that models effective strategies for asking questions and expressing concerns and needs for symptom control (i.e., pain, anxiety, depression).
* Develop Patient Narrative Videos, with women identified by their providers, to provide members of the healthcare team with a better understanding of the patient experience and issues that arise for patients outside the formal health care setting.
* Conduct a pilot test to determine whether the Patient Education Programs affect patients' experience of care, sense of control, and perceptions of caring communication, as well as knowledge, satisfaction, anxiety, depression, pain, and self-reported health.
* Determine patient and family response to Patient Narrative Videos and healthcare team response to Patient Narrative Videos and Patient Education Programs.

OUTLINE: This is a pilot, multicenter study.

A visit between the patient and his/her oncologist and healthcare team is videorecorded. Patients, family members, caregivers, and healthcare team members then undergo a 10-minute interview. Patients then undergo a 5-minute follow-up interview once every 2 weeks for 6 months. Some patients may participate in a one-time group discussion.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

PATIENT CHARACTERISTICS:

* Patients: 30 to 80 years of age
* Family members: 20 to 80 years of age
* Healthcare team members: 20 to 80 years of age
* Must be conversant in English

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Effect of Patient Education Programs on patient experience | At baseline and at 2 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Makoul, PhD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States